CLINICAL TRIAL: NCT04621942
Title: Is Inertial Training Effective and Safe Rehabilitation Method in Women After Mastectomy?
Brief Title: Inertial Rehabilitation in Women After Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University in Zielona Góra (Other)
Responsible Party: Principal Investigator, Mariusz Naczk, PhD, Head of Institute of Health Sciences, University in Zielona Góra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: University in Zielona Gora
Record Dates: First submitted 2020-10-30; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; Mastectomy; Lymphedema
Keywords: mastectomy; inertial rehabilitation; BCRL
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Intervention Model Description: the study finally included 24 women after mastectomy (age, 66.2 ± 10.6 years, range 43-82 years; body mass, 72.7 ± 10.6 kg; height, 159 ± 5.2 cm), 17 after simple mastectomy and 7 after breast conserving therapy. The participants were randomly allocated into two groups: a training group (T; n = 12) and a control group (C; n = 12) using chit method. The T group participated in 6 weeks of inertial training while the control group maintain their normal daily activity. All women still participated in rehabilitation gymnastics twice a week.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): 12 women after mastectomy. Inertial rehabilitation was performed twice a week (Monday and Thursday, between 5:00 and 8:00 PM) for 6 weeks using Cyklotren device (Inerion, Poland). Moreover, women from training group participated in rehabilitation gymnastics twice a week.
  Interventions: Other: inertial rehabilitation; Other: gymnastic rehabilitation
- Control group (Active Comparator): 12 women after mastectomy. All women participated in rehabilitation gymnastics twice a week.
  Interventions: Other: gymnastic rehabilitation

INTERVENTIONS:
Other: inertial rehabilitation — Inertial rehabilitation was performed twice a week (Monday and Thursday, between 5:00 and 8:00 PM) for 6 weeks using Cyklotren device (Inerion, Poland). Exercises were conducted by the same 2 researchers. Each training session included warm-up and 4 sets of shoulder ﬂexors, extensors, abductors, and adductors, with the right and left arms worked separately (16 sets for left and 16 sets for right arm). Each set lasted 15 seconds, a 2-minute break occurred between consecutive sets (without rest period between right and left arm). For all trained muscles 5 kg load was applied. During the training participants developed 70% of their maximal force achieved during the strength measurement. Participants observed developed during training force value displayed on-line on the screen. Cyklotren software allows to set the upper and lower limit of force; when developed strength was to low or to high a beep signal was emitted to correct participant force.
  Arms: Training group
Other: gymnastic rehabilitation — All women (from T and C group) participated in rehabilitation gymnastics twice a week during experiment (6 weeks). The gymnastics was conducted by a physiotherapist specializing in rehabilitation of women after mastectomy. The trehabilitation session lasted 45 minutes. During the sessions, the women mainly performed exercises involved shoulders, chest and the upper limbs muscles. Moreover, abdomen and back muscles were exercised.

SUMMARY:
The aim of the study was to evaluate the impact of inertial rehabilitation on: shoulder flexors, extensors and shoulder abductors and adductors strength, breast cancer-related lymphedema (BCRL) and quality of life in women after mastectomy. Twenty-four women after mastectomy were randomized to a training (T; n = 12) or control group (C; n = 12). The T group performed inertial training twice a week for 6 weeks using a Cyklotren inertial device. Each training session included warm-up and 4 sets of shoulder ﬂexors, extensors, abductors, and adductors, with the right and left arms worked. The training loads for all exercises was equal 5 kg. Before and after training the maximum force of trained muscles was tested under training conditions. Body composition, BCRL, disabilities of the arm, shoulder and hand (DASH) were also evaluated. Inertial rehabilitation caused significant improvement in strength in all tested muscles in T whereas changes in C were insignificant. Quality of life evaluated by DASH score decreased significantly in T and and did not change in C. Moreover, BCRL and body composition did not change significantly following intervention in both groups. Inertial exercises can be useful rehabilitation method in women treated for breast cancer.

DETAILED DESCRIPTION:
A group of 30 women who underwent mastectomy procedure attended an initial meeting and all of them agreed to participate in the study. The participants were members of an association of people after mastectomy (Amazons Association) and regularly participated in rehabilitation gymnastics twice a week for at least 3 years. All women met the including criteria: mastectomy was performed at least 6 months before the study, lack of: fractures in the prior 3 months, tendon and ligament injuries in the prior 2 months, serious heart disease, cerebral palsy, and limb amputations. All subjects received permission from their physician to participate in the experiment. Therefore, the study finally included 24 women after mastectomy (age, 66.2 ± 10.6 years, range 43-82 years; body mass, 72.7 ± 10.6 kg; height, 159 ± 5.2 cm), 17 after simple mastectomy and 7 after breast conserving therapy. The participants were randomly allocated into two groups: a training group (T; n = 12) and a control group (C; n = 12) using chit method. The T group participated in 6 weeks of inertial training while the control group maintain their normal daily activity. All women still participated in rehabilitation gymnastics twice a week. All participants gave written informed consent to take part in the study.

Testing

Before and after training participants were evaluated using the following tests:

* strength of shoulder muscles measurements
* body composition measurements
* breast cancer-related lymphedema (BCRL) evaluation
* disabilities of the arm, shoulder and hand test (DASH)

Strength of shoulder muscles measurement. Strength of shoulder flexors and extensors and strength of shoulder abductors and adductors were tested in the standing position using Cyklotren inertial device (Naczk 2015). After warm-up, each participant performed a 10-second maximal test of the right and left arm separately, with a 2-minute break between measurements. Participants position during strength testing and inertial training is showed on Figure1. For all measurement 5 kg load was applied. It should be noted here that the same load during inertial training doesn't mean the working muscles develop the same force. During inertial exercise force developed by muscle strongly depend on movement velocity, greater movement velocity results greater muscle load and greater force is developed (the force value is presented on-line on the Cyklotren's screen). The range of motion was approximately 90 degree (where 0 degrees corresponded to the arm along the trunk). Data collection was preceded by a familiarization session.

Body composition measurements Bioelectric impedance were used to evaluate the body composition of participants (Tanita 980 MC, Japan). The participants were asked to maintain a normal state of hydration, and they were not allowed to exercise, eat, or drink alcohol or caffeine for 12 h preceding the measurements. Measurements were conducted in the morning according to the manufacturer's guidelines. Fat mass, muscle mass, amount of water were used in future analyses.

Breast cancer-related lymphedema evaluation To evaluate the influence of inertial rehabilitation on breast cancer-related lymphedema bioimpedance spectroscopy was used. This technique allows to detect small changes in extracellular fluid (ECF) and subclinical BCRL, therefore allows for the subclinical detection of BCRL when visible swelling is not apparent. Measurements were done using L-Dex U400 unit (ImpediMed Limited, Australia). The feasibility and clinical utility of implementing L-Dex measurements in routine breast cancer care was confirmed in previous studies (Laidley and Anglin 2016, Kilgore et al 2018). During the measurements patients were lying supine on a non-metallic surface a standardized technique according to Laidley and Anglin (2016) methodology.

Disabilities of the arm, shoulder and hand test (DASH) To evaluate ability of the participants do the different daily activities DASH questionnaire was completed. DASH questionnaire is a standardized measure which captures the patients' own perspective of their upper extremity health status (Jester et. al 2005). During the questionnaire completing subjects were provided with conditions that allowed them to mark the answers freely.

Workout Inertial rehabilitation was performed twice a week (Monday and Thursday, between 5:00 and 8:00 PM) for 6 weeks using Cyklotren device (Inerion, Poland). Exercises were conducted by the same 2 researchers. Each training session included warm-up and 4 sets of shoulder ﬂexors, extensors, abductors, and adductors, with the right and left arms worked separately (16 sets for left and 16 sets for right arm). Each set lasted 15 seconds, a 2-minute break occurred between consecutive sets (without rest period between right and left arm). For all trained muscles 5 kg load was applied. During the training participants developed 70% of their maximal force achieved during the strength measurement. Participants observed developed during training force value displayed on-line on the screen. Cyklotren software allows to set the upper and lower limit of force; when developed strength was to low or to high a beep signal was emitted to correct participant force.

Statistical analysis Normality of distribution of the data was tested using the Shapiro-Wilk method. Descriptive statistics, including means and standard deviations, were calculated. For testing significance of changes analysis of variance (ANOVA) were used. The simple effect of training for each participant was defined as a relative increase in an analyzed variable after training compared with the before-training value.Lower and upper borders of 95% confidence intervals for relative increase were calculated.

Differences in relative increases between groups were tested with one-way ANOVA. If differences were detected, the Scheffé post hoc procedure was used to determine where the differences occurred. The level of significance was set at P ≤ 0.05. The effect size (ES) of the training was calculated using the paired two-sample t-test, and according to Goulet-Pelletiera and Cousineaua (2018) Cohen's d with Hedges g correction was determined. The scale presented by Cohen indicates that d < 0.41 represents a small ES, 0.41-0.70 a moderate ES, and higher than 0.70 a large ES.

ELIGIBILITY:
Inclusion Criteria:

* mastectomy performed at least 6 months before the study
* lack of fractures in the prior 3 months
* lack of tendon and ligament injuries in the prior 2 months

Exclusion Criteria:

* mastectomy was performed less than 6 months before the study
* fractures in the prior 3 months
* tendon and ligament injuries in the last 2 months
* serious heart disease
* cerebral palsy
* limb amputations

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Shoulder muscle strength | 6 weeks
  Strength of shoulder flexors and extensors and strength of shoulder abductors and adductors were tested in the standing position using Cyklotren inertial device. After warm-up, each participant performed a 10-second maximal test of the right and left arm separately, with a 2-minute break between measurements. For all measurement 5 kg load was applied. The range of motion was approximately 90 degree (where 0 degrees corresponded to the arm along the trunk). Data collection was preceded by a familiarization session.

SECONDARY OUTCOMES:
Breast cancer-related lymphedema (BCRL) | 6 weeks
  To evaluate the influence of inertial rehabilitation on breast cancer-related lymphedema bioimpedance spectroscopy was used. This technique allows to detect small changes in extracellular fluid (ECF) and subclinical BCRL, therefore allows for the subclinical detection of BCRL when visible swelling is not apparent. Measurements were done using L-Dex U400 unit (ImpediMed Limited, Australia). The feasibility and clinical utility of implementing L-Dex measurements in routine breast cancer care was confirmed in previous studies (Laidley and Anglin 2016, Kilgore et al 2018). During the measurements patients were lying supine on a non-metallic surface a standardized technique.
Disabilities of the arm, shoulder and hand test (DASH) | 6 weeks
  To evaluate ability of the participants do the different daily activities DASH questionnaire was completed. DASH questionnaire is a standardized measure which captures the patients' own perspective of their upper extremity health status (Jester et. al 2005). During the questionnaire completing subjects were provided with conditions that allowed them to mark the answers freely. The DASH test is used to assess the quality of life in women after mastectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- University in Zielona Góra, Zielona Góra, Poland

IPD SHARING:
Plan to Share IPD: No